CLINICAL TRIAL: NCT01478191
Title: Prognosis of Patients With Relapsed/Refractory Hl Treated With Combination of Ifosfamide, Gemcitabine and Vinorelbine(IGEV) Induction Therapy Before High-dose Chemotherapy (HDCT) With Autologous Hematopoietic Stem Cells Transplantation (AHSCT)
Brief Title: Prognosis of Patients With Relapsed/Refractory Hodgkin Lymphoma Treated With IGEV Induction Therapy Before HDCT With AHSCT
Acronym: IIL-ProHLRec
Status: Completed | Type: Observational
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Other Study IDs: IIL-ProHLRec; 30 (Other: AIFA)
Record Dates: First submitted 2011-10-17; First posted 2011-11-23 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2011-11

CONDITIONS: Hodgkin's Lymphoma
Keywords: Hodgkin's Lymphoma; Ifosfamide, Gemcitabine and Vinorelbine (IGEV); High Dose Chemotherapy (HDCT); Autologous Hematopoietic Stem Cells Transplantation (AHSCT)
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective analysis of a homogeneous cohort of patients with relapsed/refractory HL that received IGEV scheme as induction therapy to HDCT and AHSCT for reassess the most common prognostic factors and try to identify a prognostic score with clinical and therapeutic relevance by using 6 clinical tools:

1. B symptoms(yes/no)
2. relapse in previously irradiated areas(yes/no)
3. Ann Arbor Stage (III/IV vs I/II)
4. disease status at accrual (refractory vs relapsed)
5. Early relapse within 12 months of Complete Response (CR) versus late relapse after Complete Response (CR) lasting > l2 months",
6. extranodal involvement (yes/no).

ELIGIBILITY:
Inclusion Criteria:

* Patient with a history of classical HL relapsed/refractory which received IGEV regimen as induction therapy before high dose chemotherapy with AHSCT
* Age >18 years
* Patients with relapsed/refractory disease after standard treatments (chemotherapy +/- radiotherapy) before IGEV induction regimen. (Relapsed = disease relapse after CR.

Refractory = non CR with last chemotherapy line, or progression during last treatment, or disease progression within three months from previous treatment completion).

* Availability of clinical data, laboratory values and CT scan results of patients enrolled, performed from diagnosis to the last follow-up
* Patient scheduled to receive three or four IGEV cycles as pretransplantation induction regimen.
* First IGEV course started before December 31st 2007
* Assessment of tumor response by Cheson 1999 criteria 11

Exclusion Criteria:

* NONE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases of relapsed/refractory Hodgkin Limphoma (HL) which received full course IGEV scheme as induction therapy prior to HDCT with AHSCT from 1997 through 2007. Patients will be identified from archives of every single Center Registry database.
Sampling Method: Non-Probability Sample
Enrollment: 495 (Estimated)
Dates: Start 2010-05; Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The prognostic score will be defined taking into account Overall Survival (OS). | 4 years
  Surviving patents will be censored at the date of last known to be alive.

SECONDARY OUTCOMES:
To evaluate the defined prognostic score in terms of Progression Free Survival (PFS) | 4 years
  response rate in terms of Complete Response (CR) response rate in terms of Overall Response Rate (ORR) To validate the prognostic scores in terms of PFS and in terms OS

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, Prof., Principal Investigator — Istituto Clinico Humanitas; Monica Balzarotti, Dr., Principal Investigator — Istituto Clinico Humanitas
Locations (40):
- Italy (40):
  - Istituto Oncologico del Mediterraneo, Catania, Catania
  - Policlinico Maggiore, Milan, Italy
  - Ospedale San Gennaro, Napoli, Italy
  - Azienda Ospedaliera V. Cervello, Palermo, Italy
  - Azienda Ospedaliera "Bianchi Melacrino Morelli", Reggio Calabria, Italy
  - Presidio Ospedaliero - Unità Complessa Ematologia, Treviso, Italy
  - Ematologia e Trapianto IRCCS, Istituto Nazionale dei Tumori, Milan, Milano
  - SCDU Ematologia, AOU Maggiore della Carità, Novara, Novara
  - Ospedale dell'Angelo, Mestre, VE
  - A.O.SS. Biagio, Antonio e Cesare Arrigo, Alessandria
  - AORN San G.Moscati, Avellino
  - Centro di riferimento Oncologico - Oncologia Medica A, Aviano (PN)
  - Divisione di Ematologia Spedali Civili, Brescia
  - Ospedale di Circolo, Busto Arsizio - VA
  - Divisione di Ematologia Osp.Businco, Cagliari
  - Ospedale civile Divisione di Ematologia, Civitanova Marche (MC)
  - Ospedale S Martino, Genova
  - Ospedale San Martino - Divisione di Ematologia, Genova
  - Ospedale Santa Maria Goretti, Latina
  - A O Papardo, Messina
  - Azienda Ospedaliero Universitaria Policlinico Gaetano Martino, Messina
  - Osp. San Carlo Borromeo Divisione di Oncologia Medica, Milan
  - Ospedale Niguarda CA' Granda, Milan
  - Policlinico di Modena - Università degli studi, Modena
  - AOU Federico II di Napoli, Napoli
  - Ospedale Umberto I UO Med. Interna Oncoematologia, Nocera Inferiore (SA)
  - A.O. di Padova Divisione di Oncologia Medica, Padua
  - Policlinico P.Giaccone, Palermo
  - Fondazione Policlinico San Matteo, Pavia
  - Ospedale Santo Spirito Dipartimento di Ematologia, Pescara
  - Ospedale Civile G.da Saliceto - UOA Ematologia, Piacenza
  - AO Santa Maria Nuova, Reggio Emilia
  - Ospedale Oncologico regionale CROB, Rionero in Vulture (PZ)
  - Ospedale S. Eugenio, Roma
  - Policlinico Università Tor Vergata, Roma
  - Univeristà La Sapienza, Roma
  - Clinica Humanitas, Rozzano (MI)
  - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo (FG)
  - Istituto di Ematologia Università degli studi di Sassari, Sassari
  - Ematologia II OspedaleSan Giovanni Battista Molinette, Torino